CLINICAL TRIAL: NCT06416774
Title: A Phase I Clinical Study to Evaluate the Safety, Biodistribution, Radiation Dose and Pharmacokinetics of 68Ga-HX01 Injection for PET Imaging
Brief Title: A Clinical Study of 68Ga-HX01 Injection for PET Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hexin (Suzhou) Pharmaceutical Technology Co., Ltd (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0688
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Malignancy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ia: Low-dose group (Experimental): The injection dose of 68Ga-HX01 for low-dose group is 0.05 mCi/kg.
  Interventions: Drug: 68Ga-HX01 Injection(0.05mCi/kg)
- Ia: High-dose group. (Experimental): The injection dose of 68Ga-HX01 for the high-dose group is 0.1 mCi/kg.
  Interventions: Drug: 68Ga-HX01 Injection(0.1mCi/kg)
- Ib: Patients with malignancy. (Experimental): The injection dose for phase Ib patients was 0.07 mCi/ kg.
  Interventions: Drug: 68Ga-HX01 Injection(0.07mCi/kg)

INTERVENTIONS:
Drug: 68Ga-HX01 Injection(0.05mCi/kg) — The study is divided into three stages, including screening period, administration period and follow-up observation period. The maximum screening period is 7 days. Eligible subjects will receive intravenous injection of the experimental drug 68Ga-HX01 on Day 1 of the study and undergo PET imaging, while blood and urine are collected for radioactive counts for pharmacokinetic analysis and safety monitoring.
  They will return to the study center for safety checks on Day 2 after injection and phone follow-up on Day 7 for adverse events and drug combinations/treatments.
  Other Names: 68Ga-HX01
  Arms: Ia: Low-dose group
Drug: 68Ga-HX01 Injection(0.1mCi/kg) — The study is divided into three stages, including screening period, administration period and follow-up observation period. The maximum screening period is 7 days. Eligible subjects will receive intravenous injection of the experimental drug 68Ga-HX01 on Day 1 of the study and undergo PET imaging, while blood and urine are collected for radioactive counts for pharmacokinetic analysis and safety monitoring.
  They will return to the study center for safety checks on Day 2 after injection and phone follow-up on Day 7 for adverse events and drug combinations/treatments.
  Other Names: 68Ga-HX01
  Arms: Ia: High-dose group.
Drug: 68Ga-HX01 Injection(0.07mCi/kg) — The study is divided into three stages, including screening period, administration period and follow-up observation period. The maximum screening period is 7 days. Eligible subjects will receive intravenous injection of the experimental drug 68Ga-HX01 on Day 1 of the study and undergo PET imaging, while blood and urine are collected for safety monitoring.
  They will return to the study center for safety checks on Day 2 after injection and phone follow-up on Day 7 for adverse events and drug combinations/treatments.
  Other Names: 68Ga-HX01
  Arms: Ib: Patients with malignancy.

SUMMARY:
This is a single-center, open Phase I clinical study, consisting of two parts: a Phase Ia study in healthy adult subjects and a Phase Ib study in patients with malignant solid tumors.

DETAILED DESCRIPTION:
Phase Ia design:

The Phase Ia study is designed to evaluate the safety, biodistribution (PET imaging), radiation dose, and pharmacokinetics of 68Ga-HX01 injection after a single intravenous administration in healthy Chinese adult subjects.

Twelve healthy adult subjects will be enrolled in the Phase Ia program.

Phase Ib design:

The purpose of the Phase Ib clinical study is to evaluate the safety and biodistribution (PET imaging) of patients with malignant solid tumors receiving a single intravenous administration of 68Ga-HX01 injection, and to explore the characteristics of tumor imaging.

Ten patients with malignant solid tumors will be enrolled in Phase Ib.

ELIGIBILITY:
This study consists of two parts: a Phase Ia study in healthy adult subjects and a Phase Ib study in patients with malignant solid tumors.

Phase Ia:

Inclusion Criteria:

* 18-50 years old;
* Female weight 45-80kg, male weight 50-80kg;
* Agree to take effective contraception during the study and for at least three months after the drug administration.

Exclusion Criteria:

* Pregnant or lactating women; Or plan to donate sperm or eggs during the study or within three months after drug administration;
* Known or suspected allergic to the test drug or any of its components;
* Receiving another investigational drug at the time of enrollment, or within 5 half-lives of the drug at the time of enrollment;
* Those who tested positive for hepatitis B/C virus, syphilis or HIV during screening;
* Clinically significant abnormalities in hematology, blood biochemistry, and urine routine during screening;
* Patients with clinically significant diseases within 4 weeks before screening;
* Blood pressure higher than 150/100 mmHg or lower than 90/50 mmHg at screening;
* Use of any prescription or over-the-counter drugs within 2 weeks before the trial drug administration;
* Blood donation or blood loss ≥500 mL within 12 weeks before administration;
* History of drug or alcohol abuse within 12 months prior to administration;
* Smoking more than 5 cigarettes a day or consuming the same amount of nicotine or nicotine replacement within 3 months before administration;
* History of malignancy;
* Plan to schedule surgery and other invasive interventions within one week of the test drug injection;
* Compliance to lie for about 90 minutes during the PET examination.

Phase Ib:

Inclusion Criteria:

* Patients with malignant solid tumors with measurable lesions (target lesions) confirmed by histopathology or cytology or clinical diagnosis;
* 18-75 years old;
* Eastern Cooperative Oncology Group (ECOG) score 0 or 1;
* life expectancy ≥6 months;
* Agree to take effective contraception during the study and for at least three months after the drug administration.

Exclusion Criteria:

* Pregnant or lactating women; Or plan to donate sperm or eggs during the study or within three months after drug administration;
* Known or suspected allergic to the test drug or any of its components;
* Receiving another investigational drug at the time of enrollment, or within 5 half-lives of the drug at the time of enrollment;
* Those who tested positive for hepatitis B/C virus, syphilis or HIV during screening;
* Any radiotherapeutic drugs used within 90 days before administration, or any radionuclide diagnostic drugs received within 3 days before administration;
* Plan to schedule surgery and other invasive interventions within 2 days after trial drug injection;
* Abnormal liver and kidney function: serum total bilirubin (TBIL) > 1.5×ULN (upper limit of normal), or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5×ULN, or serum creatinine > 1.5×ULN;
* With active infection at the time of screening;
* Compliance to lie for about 60 minutes during the PET examination.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Temperature | During the screening period (within 7 days), within 30 minutes before 68Ga-HX01 administration, 1.0 to 1.5 hours, 3.0 to 3.5 hours after the injection and Day 2.
  Changes in body temperature after 68Ga-HX01 administration were recorded to analyze the effects of 68Ga-HX01 on body temperature.
Respiration | Time Frame: During the screening period, within 30 minutes before 68Ga-HX01 administration, 1.0 to 1.5 hours, 3.0 to 3.5 hours after the injection and Day 2.
  Changes in respiration rate after 68Ga-HX01 administration were recorded to analyze the effects of 68Ga-HX01 on respiration.
Pulse | During the screening period, within 30 minutes before 68Ga-HX01 administration, 1.0 to 1.5 hours, 3.0 to 3.5 hours after the injection and Day 2.
  Changes in pulse after 68Ga-HX01 administration were recorded to analyze the effects of 68Ga-HX01 on pulse.
Blood pressure | During the screening period, within 30 minutes before 68Ga-HX01 administration, 1.0 to 1.5 hours, 3.0 to 3.5 hours after the injection and Day 2.
  Changes in diastolic pressure and systolic pressure after 68Ga-HX01 administration were recorded to analyze the effects of 68Ga-HX01 on blood pressure.
Oxygen saturation | During the screening period, within 30 minutes before 68Ga-HX01 administration, 1.0 to 1.5 hours, 3.0 to 3.5 hours after the injection and Day 2.
  Changes in oxygen saturation after 68Ga-HX01 administration were recorded to analyze the effects of 68Ga-HX01 on oxygen saturation.
Electrocardiogram QT Interval | Within 30 minutes before 68Ga-HX01 administration, 3.0 to 3.5 hours after the injection and Day 2.
  Electrocardiogram QT interval was recorded to assess the effect of 68Ga-HX01 administration.
Electrocardiogram QRS Interval | Within 30 minutes before 68Ga-HX01 administration, 3.0 to 3.5 hours after the injection and Day 2.
  Electrocardiogram QRS interval was recorded to assess the effect of 68Ga-HX01 administration.
Electrocardiogram PR Interval | Within 30 minutes before 68Ga-HX01 administration, 3.0 to 3.5 hours after the injection and Day 2.
  Electrocardiogram PR interval was recorded to assess the effect of 68Ga-HX01 administration.
Electrocardiogram T Wave | Within 30 minutes before 68Ga-HX01 administration, 3.0 to 3.5 hours after the injection and Day 2.
  The shape of electrocardiogram T wave was recorded to assess the effect of 68Ga-HX01 administration.
Electrocardiogram ST Segment | Within 30 minutes before 68Ga-HX01 administration, 3.0 to 3.5 hours after the injection and Day 2.
  The shape of electrocardiogram ST segment was recorded to assess the effect of 68Ga-HX01 administration.
Number of Participants With Abnormal Laboratory Values in Blood routine | Day 2.
  The blood routine of Day 2 was recorded.
Number of Participants With Abnormal Laboratory Values in Blood biochemistry | Day 2.
  Blood biochemistry of Day 2 was recorded.
Prothrombin time test and/or a partial thromboplastin time test (PTT) | Day 2.
  Coagulation function of Day 2 was recorded.
Number of Participants With Abnormal Laboratory Values in Urine routine | Day 2.
  Urine routine of Day 2 was recorded.

SECONDARY OUTCOMES:
Dosimetry | At 10, 30, 60 and 120 minutes after 68Ga-HX01 injection.
  OLINDA/EXM software was used to calculate the radiation dose using the uptake of each organ and tissue in Ia subjects. The uptake values are calculated from the SUV values of PET images at each time point.
The percentage of injected dose per gram (% ID/g) | Blood samples are collected for the radioactivity determination before (within 30 minutes) and after 68Ga-HX01 injection at different time points (2, 5, 10, 30, 60, 90, 120, and 180 minutes).
  The blood radioactivity time-activity curve was drawn based on the percentage of injected dose per gram (% ID/g) of blood samples at each time point.
The max uptake of each lesion | At 30 and 60 minutes after 68Ga-HX01 injection.
  SUVmax was automatically calculated to quantify 68Ga-HX01 uptake in the lesions.
The mean uptake of each lesion | At 30 and 60 minutes after 68Ga-HX01 injection.
  SUVmean was automatically calculated to quantify 68Ga-HX01 uptake in the lesions.
Lesion number | At 30 and 60 minutes after 68Ga-HX01 injection.
  Lesion number was recorded.
The size of each lesion | At 30 and 60 minutes after 68Ga-HX01 injection.
  Lesion size was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Gai Y, Ye T, Fan L, Xiu L, Ruan W, Hu F, Chen J, Lan X. Head-to-head evaluation of [18F]FDG PET/CT and [68Ga]Ga-HX01 PET/MR in sarcoma patients. Eur J Nucl Med Mol Imaging. 2025 Jul;52(8):2898-2905. doi: 10.1007/s00259-025-07130-4. Epub 2025 Feb 20. PMID 39976700
- [Derived] Zhang X, Fang H, Yang B, Qin C, Hu F, Ruan W, Chen J, Zeng D, Gai Y, Lan X. Phase I study of [68Ga]Ga-HX01 for targeting integrin alphavbeta3 and CD13 in healthy and malignancy subjects. Eur J Nucl Med Mol Imaging. 2025 Mar;52(4):1293-1304. doi: 10.1007/s00259-024-07002-3. Epub 2024 Nov 29. PMID 39609274